CLINICAL TRIAL: NCT06162065
Title: Effectiveness of Oral Boldo in Improving Urinary Symptoms and Body Stability in Women Diagnosed With Overactive Bladder
Brief Title: Effectiveness of Oral Boldo in Women With Overactive Bladder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Uro Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118/2023
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urinary, Overactive Bladder, Boldine
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — oxybutynin

STUDY DESIGN:
Intervention Model Description: prospective experimental study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): women with overactive bladder will be treated using oral antimuscarinics for 4 weeks under strict medical indication, with a treatment scheme consisting of 10 mg tablet of oxybutynin once a day.
  Interventions: Drug: Oxybutynin Pill
- Group 2 (Experimental): 5 women will receive combined oral treatment. 1 tablet of 10 mg once a day of oral of oxybutynin and they will also be supplemented with powder boldo capsules for 4 weeks under strict medical indication. This group will be supplemented with 1 capsules of 340 mg every 8 hours of boldo (take suggested by the manufacturer), for 5 days in a row and 5 days off.
  Interventions: Drug: Oxybutynin Pill; Dietary Supplement: Boldo supplement

INTERVENTIONS:
Drug: Oxybutynin Pill — pharmacological antimuscarinic treatment
Dietary Supplement: Boldo supplement — treatment supplemented with boldo
  Arms: Group 2

SUMMARY:
The objective of this clinical trial is to know if boldo oral powder capsules works well in the management of urinary symptoms in women with overactive bladder. The main questions it aims to answer are:

* Is boldo supplementation safe?
* Does boldo improve urinary parameters and body stability? 5 participants will be treated with an oral antimuscarinic (oxybutynin) and supplemented with oral spray bolus. The urinary chart will be applied to measure urinary frequency and voiding intervals. In addition, urinary symptoms and the level of discomfort they generate will be measured. Finally, the MiniBest test will be applied using a portable device which acts as an inertial sensor to record the movements made. For comparative purposes, 5 women who will only be treated with the oral antimuscarinic (oxybutynin) will be measured to see if there are significant differences between the medication alone versus the supplemented medication.

DETAILED DESCRIPTION:
10 women over 18 years of age who meet the selectivity criteria will be recruited under written informed consent, previously approved by the competent ethics committee. Patients will be diagnosed with overactive bladder through a clinical interview and a voiding record performed by a specialist urologist that may or may not be confirmed by a urodynamic study.

Prior to carrying out the tests, the informed consent will be read aloud to the patient by one of the responsible researchers, explaining the relevant aspects and any doubts that may arise in this regard. The document must be signed by each recruited patient if she wishes to participate voluntarily.

Additionally, your vital signs will be assessed to ensure your safety when taking measurements and baseline data will be generated. The self-application of the voiding chart will be explained to them, which should be done once a week throughout the treatment.

A postural evaluation through a stability test will be performed on all patients using a portable device placed through a harness. The cell phone has inertial sensors and will record position signals. This measurement will be carried out in two instances: pre-intervention and post-intervention to obtain postural parameters of anticipatory adjustments, reactive strategies, sensory orientation and dynamic gait.

Subsequently, the total sample will be randomly subdivided into two groups consisting of 5 patients. The first group will be treated through the use of oral antimuscarinics for 4 weeks under strict medical indication, with a treatment scheme consisting of 10 mg oxybutynin tablet once a day, while the other 5 remaining subjects will receive a combined oral treatment using the use of oral antimuscarinic under the same scheme (10 mg oxybutynin tablet once a day), but they will also be complemented with boldo powder for 4 weeks under strict medical indication. This last group will be complemented with 1 capsules of 380 mg every 8 hours of boldo (take suggested by the manufacturer), for 5 days in a row and 5 days off.

Patients will be monitored weekly by telephone and asked to report the results of the self-administered voiding record while the bladder control questionnaire for overactive bladder symptoms is administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with urinary urgency, frequency, nocturia, with or without urgency urinary incontinence.

Exclusion Criteria:

* Excessive fluid intake. Use of diuretics. Neurological diseases or cognitive impairment (e.g., stroke, multiple sclerosis, spinal cord injury), mobility deficits, medically complicated/uncontrolled diabetes, fecal motility disorders (fecal incontinence/constipation), chronic pelvic pain, history of recurrent urinary tract infections (UTI), gross hematuria, previous pelvic/vaginal surgeries (incontinence/prolapse surgeries), pelvic cancer (bladder, colon, cervix, uterus, prostate), pelvic radiation, female patient with significant prolapse (GIII and IV), pelvic floor disorders (e.g., spasticity of the pelvic floor muscles, pain or any pathology that could appear overactive bladder masking other diagnoses, glaucoma, drug or supplement allergy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms | 1 month
  Using a urinary chart, measure urinary frequency and intervals.
Bladder Control Self-Assessment Questionnaire | 1 month
  measure the presence of urinary urgency and urine leakage along with the level of discomfort this produces
MiniBESTest | 1 month
  Balance systems evaluation test (anticipatory, reactive postural control, sensory orientation, dynamic gait)

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Uromed, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gibson W, Jones A, Hunter K, Wagg A. Urinary urgency acts as a source of divided attention leading to changes in gait in older adults with overactive bladder. PLoS One. 2021 Oct 4;16(10):e0257506. doi: 10.1371/journal.pone.0257506. eCollection 2021. PMID 34606514
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Neuhaus J, Pfeiffer F, Wolburg H, Horn LC, Dorschner W. Alterations in connexin expression in the bladder of patients with urge symptoms. BJU Int. 2005 Sep;96(4):670-6. doi: 10.1111/j.1464-410X.2005.05703.x. PMID 16104929
- [Background] Subedi YP, Altenberg GA, Chang CT. Advances in the development of connexin hemichannel inhibitors selective toward Cx43. Future Med Chem. 2021 Feb;13(4):379-392. doi: 10.4155/fmc-2020-0291. Epub 2021 Jan 5. PMID 33399487
- [Background] Cea LA, Vasquez W, Hernandez-Salinas R, Vielma AZ, Castillo-Ruiz M, Velarde V, Salgado M, Saez JC. Skeletal Muscle Atrophy Induced by Diabetes Is Mediated by Non-Selective Channels and Prevented by Boldine. Biomolecules. 2023 Apr 21;13(4):708. doi: 10.3390/biom13040708. PMID 37189454
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Nowakowski L, Kulik-Rechberger B, Wrobel A, Rechberger T. [Overactive bladder--a new insight into the pathogenesis of its idiopathic form]. Ginekol Pol. 2012 Nov;83(11):844-8. Polish. PMID 23379193
- [Background] Christ GJ, Day NS, Day M, Zhao W, Persson K, Pandita RK, Andersson KE. Increased connexin43-mediated intercellular communication in a rat model of bladder overactivity in vivo. Am J Physiol Regul Integr Comp Physiol. 2003 May;284(5):R1241-8. doi: 10.1152/ajpregu.00030.2002. PMID 12676745
- [Background] Ikeda Y, Fry C, Hayashi F, Stolz D, Griffiths D, Kanai A. Role of gap junctions in spontaneous activity of the rat bladder. Am J Physiol Renal Physiol. 2007 Oct;293(4):F1018-25. doi: 10.1152/ajprenal.00183.2007. Epub 2007 Jun 20. PMID 17581924
- [Background] Backhouse N, Delporte C, Givernau M, Cassels BK, Valenzuela A, Speisky H. Anti-inflammatory and antipyretic effects of boldine. Agents Actions. 1994 Oct;42(3-4):114-7. doi: 10.1007/BF01983475. PMID 7879695
- [Background] O'Brien P, Carrasco-Pozo C, Speisky H. Boldine and its antioxidant or health-promoting properties. Chem Biol Interact. 2006 Jan 5;159(1):1-17. doi: 10.1016/j.cbi.2005.09.002. Epub 2005 Oct 10. PMID 16221469
- [Background] Gotteland M, Espinoza J, Cassels B, Speisky H. [Effect of a dry boldo extract on oro-cecal intestinal transit in healthy volunteers]. Rev Med Chil. 1995 Aug;123(8):955-60. Spanish. PMID 8657963
- [Background] Peng B, Xu C, Wang S, Zhang Y, Li W. The Role of Connexin Hemichannels in Inflammatory Diseases. Biology (Basel). 2022 Feb 2;11(2):237. doi: 10.3390/biology11020237. PMID 35205103
- [Background] Booth J, Paul L, Rafferty D, Macinnes C. The relationship between urinary bladder control and gait in women. Neurourol Urodyn. 2013 Jan;32(1):43-7. doi: 10.1002/nau.22272. Epub 2012 Jun 12. PMID 22693146